CLINICAL TRIAL: NCT06231498
Title: Disease Susceptibility and Response to IL5 Blockade in Patients With Eosinophilic Granulomatosis With Polyangiitis (EGPA): an Epigenome-wide Association Study Integrated With Transcriptomic and Proteomic Analyses
Brief Title: The Epigenomic Signature of Eosinophilic Granulomatosis With Polyangiitis
Acronym: EPI-EGPA
Status: Not yet recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Careggi Hospital (Other); University of Florence (Other)
Responsible Party: Principal Investigator, Augusto Vaglio, Professor, Meyer Children's Hospital IRCCS
Other Study IDs: EPI-EGPA
Record Dates: First submitted 2023-11-14; First posted 2024-01-30 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis
Keywords: Epigenome; DNA Methylation; Eosinophilic Granulomatosis with Polyangiitis; EGPA
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A peripheral whole blood sample for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overall Cohort: The study will include 300 adult (>18yo) patients with Eosinophilic Granulomatosis with Polyangiitis (EGPA). All patients will be recruited at Meyer Children's Hospital and Careggi University Hospital, which are referral centers for EGPA and have a large cohort of prevalent cases under long-term follow-up. They will represent the cases for the case-control epigenome-wide association study. Patients are expected to be untreated or under glucocorticoids at the time of sampling. A blood sample will be drawn for each participant. Among this cohort, 50 patients will be identified that will undergo treatment with Mepolizumab, and they will form the sub-cohort in which we will search for epigenetic predictors of the response to Mepolizumab treatment (predictive epigenomic study). These 50 patients will also be analyzed with regard to the transcriptomic and proteomic profile. Written informed consent from all participants and approval from the local ethical committees will be obtained.

SUMMARY:
This is a case-control observational study on blood samples. The primary goal of this study is to identify the epigenetic marks that can distinguish patients suffering from Eosinophilic Granulomatosis with Polyangiitis (EGPA) from healthy individuals. The secondary goal is to identify epigenetic or transcriptional marks that can predict if a patient with EGPA will benefit from therapy with Mepolizumab. This study is observational, meaning there will be no alterations of patients' routine clinical care. A blood sample will be drawn for each patient. If the patient will undergo treatment with Mepolizumab (based on routine clinical care), then the blood sample will be drawn before Mepolizumab initiation. The blood samples will be used for genome-wide DNA methylation profiling and for transcriptomic profiling. Healthy individuals as controls for the association study will not be recruited. In fact, the epigenetic and transcriptomic data obtained from EGPA patient blood will be compared against already available genome-wide DNA methylation and transcriptomic profiles of the blood of healthy individuals from previous studies. A total of 300 patients with EGPA will be recruited for the study. The first part of the study, corresponding to the primary goal, will involve all of the 300 patients. The second part of the study, corresponding to the secondary goal, will involve a study population subset consisting of 50 patients.

DETAILED DESCRIPTION:
Background and Rationale. Eosinophilic Granulomatosis with Polyangiitis (EGPA) is a rare multisystem immune-mediated disease classified both among Anti Neutrophil Cytoplasmic Antibody (ANCA)-associated vasculitis and among hypereosinophilic disorders. Current scientific knowledge describes EGPA as a complex or multifactorial nature of the disease, i.e. the disease is triggered by a combination of inherited genetic variants and environmental factors. The term "epigenetics" refers to heritable alterations in gene expression which do not correspond to a variation in the underlying DNA sequence. In the context of various autoimmune diseases similar to EGPA and in the context of asthma (a condition that almost all EGPA patients suffer from), several studies have highlighted that epigenetics plays a fundamental role in the pathogenesis/pathophysiology and that in particular it can potentially represent the mechanism by which environmental exposures interact with genetics to cause the disease. Therefore, studying epigenetics (and namely DNA methylation as the most studied epigenetic mechanism) in EGPA could lead to an in-depth knowledge of the pathology and in particular to the identification of epigenetic markers, useful in diagnosis, or in monitoring disease activity, or in predicting response to pharmacological treatment.

Objectives. The primary objective is the identification of loci whose methylation level is associated with the pathology (i.e. epigenetic markers of the disease). The secondary objectives are: identification of loci whose methylation level correlates with the response to treatment with the drug Mepolizumab in patients affected by the disease (i.e. epigenetic markers predictive of response to Mepolizumab); identification of genes whose transcription level is related to the disease and of proteins whose plasma concentration is related to the disease (in this way, we expect to evaluate the effects of epigenetic variation on gene/protein expression and to identify the corresponding biological pathways); identification of epigenetic predictors of disease outcomes, e.g. remission, relapse, survival; identification of epigenetic markers of the main disease subphenotypes, i.e. the ANCA+ and ANCA- subsets.

Study Design. Observational case-control study on biological samples. The study is divided into two different parts: The first part is a genome-wide DNA methylation case-control association study. The genome-wide methylation profile derived from blood samples from 300 patients will be compared to the methylation profile in the blood of healthy individuals. The second part is a predictive study, aiming at assessing whether epigenetics can be used to predict the response to Mepolizumab. This part of the study will cover a study population subset, consisting of 50 patients who will undergo treatment with Mepolizumab (as part of their clinical routine) and whose blood sample will be drawn before starting Mepolizumab therapy. Not only the genome-wide methylation profile will be obtained from the blood (like all the other patients included in the study), but also the transcriptomic profile. These profiles will be analyzed to search for loci whose level of methylation and/or expression correlate with the response to treatment with Mepolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who meet the 1990 American College of Rheumatology classiﬁcation criteria for EGPA or the criteria proposed in the MIRRA trial, or the 2022 American College of Rheumatology/European Alliance of Associations for Rheumatology classification criteria;
* Written informed consent from all the study participants.

Exclusion Criteria:

* Patients with inadequate or unavailable data regarding response to treatment at months 6 and 12 after Mepolizumab initiation will be included in the case-control Epigenome-Wide Association Study (EWAS) but not in the predictive epigenomic study;
* Patients with childhood-onset EGPA;
* Patients who are pregnant or breast-feeding.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 300 adult (>18yo) patients with Eosinophilic Granulomatosis with Polyangiitis (EGPA). All patients will be recruited at Meyer Children's Hospital and Careggi University Hospital, which are referral centres for EGPA and have a large cohort of prevalent cases under long-term follow-up. They will represent the cases for the case-control epigenome-wide association study. Patients are expected to be untreated or under glucocorticoids at the time of sampling. A blood sample will be drawn for each participant. Among this cohort, 50 patients will be identified that will undergo treatment with Mepolizumab, and they will form the sub-cohort in which epigenetic predictors of the response to Mepolizumab treatment (predictive epigenomic study) will be searched for.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Epigenome-Wide Association Study | Through study completion, an average of 1 year
  The primary objective of the study is the identification of loci whose methylation level is associated with the pathology (i.e. epigenetic markers of the disease). This means that there is not any outcome that will be measured with regard to the primary objective.
Mepolizumab Therapy Response | 6 months and 12 months after Mepolizumab therapy initiation
  The main secondary objective of the study is the identification of loci whose methylation level correlates with the response to treatment with the Mepolizumab in patients with EGPA (i.e. epigenetic predictors of response to Mepolizumab). To this end, the response to treatment with Mepolizumab is the outcome that will be measured. Complete response to treatment will be deﬁned as no disease activity (Birmingham Vasculitis Activity Score = 0) and a prednisolone or prednisone dose (or equivalent) of ≤4.0 mg/day, as deﬁned by the MIRRA trial. Partial response to treatment will be deﬁned as no disease activity and a prednisone dose (or equivalent) of >4.0 mg/day.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Vaglio, MD, PhD, Principal Investigator — Meyer Children's Hospital IRCCS

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers other than the study investigators